CLINICAL TRIAL: NCT06961877
Title: Talking About Cannabis: Developing an Intervention for Family Members of Young Adults With FEP to Support Reduced Cannabis Use
Brief Title: Skills for Talking About Cannabis for Families of Young Adults With Psychosis
Acronym: STAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denise Walker, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022601; 1R34MH133684-01A1 (NIH)
Record Dates: First submitted 2025-04-24; First posted 2025-05-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Caregiver Burden; Cannabis Use; Expressed Emotion; Communications Skills
Keywords: coordinated specialty care; cannabis use disorder; first episode psychosis; caregiver burden; cannabis use; communication skills
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis Conversation Skills for Families (CCSF) (Experimental): The purpose of the intervention is to train family members in communication skills that may increase contemplation of change in their loved one with first episode psychosis to reduce cannabis use, decrease conflict surrounding these discussions, and provide skills to understand when and how to approach their loved one about cannabis use and encourage treatment.
  Six sessions (90 minutes each) will be held weekly in a closed group format via Zoom, with the same therapist leading each group. Group size will be 3-8 participants, with an average wait time of 4 weeks. Assessments will occur at baseline, post-treatment, and at a 3-month follow-up.
  Interventions: Behavioral: Cannabis Conversation Skills for Families (CCSF)
- Treatment as Usual (TAU) Control (No Intervention): In this project, treatment as usual will consist of psychoeducation on cannabis and its impacts on psychosis and family services otherwise provided to participants through their participation in the coordinated specialty care program at which their loved one is enrolled. The investigators will track what each family receives and characterize the content and dose in analysis.

INTERVENTIONS:
Behavioral: Cannabis Conversation Skills for Families (CCSF) — The purpose of the intervention is to train family members in communication skills that may increase contemplation of change in their loved one with first episode psychosis to reduce cannabis use, decrease conflict surrounding these discussions, and provide skills to understand when and how to approach their loved one about cannabis use and encourage treatment. Because families report confusion from the mixed messages they receive about cannabis and also desire research-based information, CCSF will involve psychoeducation on the risks and relationship of cannabis to psychosis to increase participants motivation to engage in the intervention. frequency of cannabis use as it relates to psychosis treatment outcomes.
  Arms: Cannabis Conversation Skills for Families (CCSF)

SUMMARY:
The objectives of this research is to (1) create a family intervention and provider manual to train family members of young people with psychosis (YP-P) who are heavy cannabis users new communication skills to motivate change in the YP-P's cannabis use, (2) pre-test the intervention with 10 family member participants and adapt the intervention based on their recommendations, and (3) evaluate the feasibility and acceptability of the intervention in a randomized pilot trial (n=40). The investigators anticipate that the intervention will improve family participants' communication skills, decrease expressed emotion and caregiver burden. The investigators anticipate that improvements in communication skills, expressed emotion and caregiver burden will lead to decreases in the cannabis use of their YP-P.

DETAILED DESCRIPTION:
The objectives of this research will be implemented in two phases. Phase II will develop a family intervention informed by a Stakeholder Advisory Board and pre-test the intervention will be adapted with 10 family member participants. The intervention based on recommendations in phase 1. The investigators anticipate that the intervention will improve family participants' communication skills, decrease expressed emotion and caregiver burden. The investigators anticipate that improvements in communication skills, expressed emotion and caregiver burden will lead to decreases in the cannabis use of their YP-P.

Phase 2 will evaluate the acceptability, feasibility, and preliminary effect sizes of the intervention in a pilot randomized controlled trial comparing it to treatment as usual (TAU) with 40 family participants. This pilot test is consistent with the stated purpose of Stage 1B of the NIH Stage Model for behavioral intervention development and the R34 mechanism of "providing resources for evaluating the feasibility, tolerability, acceptability and safety and preliminary effectiveness of approaches to improve mental health/functional outcomes". The purpose of this pilot study is to develop and test the feasibility and acceptability of the intervention protocol, study procedures, and recruitment plan. Secondarily, the investigators intend to collect data to inform effect size estimates on outcomes to plan for an R01.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older,
2. has a loved one who is both in CSC treatment for FEP and has used cannabis in the past 30 days,
3. has regular contact with their loved one with FEP. It is assumed that YA-P will be aged 13-40 with schizophrenia spectrum disorder given criteria for CSC enrollment.

Exclusion Criteria:

1. Unable to read study materials and communicate feedback in English
2. Do not have access to Zoom

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Cannabis and psychosis knowledge | baseline, 3 month follow-up
  Cannabis knowledge test. This measure does not use a scale; multiple choice items test understanding of cannabis products, consumption, and impacts. Higher scores indicate higher level of cannabis knowledge.
Caregiver Burden Index | baseline, 3 month follow-up
  The CBI is a 24-item assessment of both objective (time away from work for caregiving) and subjective (psychological impact) burden of caregiving in a Likert-format scale (0-4) that measures five dimensions of caregiver burden: time dependence, developmental, physical, social, and emotional burden. Each sub scale ranges from 0 (low ) to 20 (high).
Family Attitudes Scale (FAS) | baseline, 3 month follow-up
  The FAS is a 30-item self-report measure of expressed emotion (EE) using a Likert scale (e.g., 1 to 5); higher scores indicate more positive attitudes towards family dynamics, while lower scores suggests negative attitudes.
Timeline Followback - Collateral version (TLFB-C) | baseline, 3 month follow up
  The TLFB will ask participants to complete a calendar for the past 30 days indicating the days they believe their YA-P used cannabis and other substances.
Motivational Interviewing Treatment Integrity (MITI) | baseline, post-treatment (6 week)
  Participants will complete an audio-recorded encounter with a standardized patient who will remain in character as a YA-P who uses cannabis.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 3 month follow up
  Intervention satisfaction will be assessed with the CSQ-8, a widely used instrument, consisting of eight items each answered on a 4-point scale. The possible scores range from 8 to 32, with higher scores indicating a greater level of overall satisfaction with the services received.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Walker, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- The University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All scientific data (survey response data) will be both preserved and shared. Data will be made publicly available to the research community. This will include but may not be limited to (a) survey items and corresponding response options (including missingness coding), (b) a codebook for scoring survey items and composite scales, (c) a detailed description of internally computed variables (e.g., time spent viewing intervention content), and (d) documentation of intervention components that participants were exposed to (both treatment and control conditions). Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the NIAAA Data Archive.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be shared with the general research community at the time of an associated publication, or the end of the award/support period, whichever comes first.
Access Criteria: The data will be made available for sharing with the general research community via the NDA website. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NDA data by submitting a data access request in accordance with applicable NDA policies.